CLINICAL TRIAL: NCT00165009
Title: A Prospective Randomized Comparison of a Novel Hemostatic Clip (Resolution Clip™) to Combined Epinephrine Injection and Heater Probe Thermocoagulation in the Endoscopic Control of Ulcer Bleeding
Brief Title: Resolution Endoclips Vs Epinephrine Injection and Heater Probe
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RET
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: Bleeding Peptic Ulcer; Endoscopic treatment
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DUAL THERAPY (No Intervention): DUAL THERAPY
- 'Resolution clip (Experimental): 'Resolution clip
  Interventions: Device: Resolution clip (endo-clipping device)

INTERVENTIONS:
Device: Resolution clip (endo-clipping device) — Resolution clip (endo-clipping device)
  Arms: 'Resolution clip

SUMMARY:
To compare the efficacy of a novel endoscopic clipping device(Resolution Clip™) and conventional epinephrine injection and heater probe thermocoagulation in control of peptic ulcer bleeding and prevention of recurrent bleeding

DETAILED DESCRIPTION:
The mortality of peptic ulcer bleeding remains high despite advances in endoscopy and medical therapy. Endoscopic therapy effectively controls peptic ulcer bleeding and substantially reduces recurrent bleeding. However, the best endoscopic therapy is still unclear. The current standard of therapy is injection with diluted epinephrine and heater probe (3.2mm) thermo-coagulation. However, it may be associated with complications such as precipitation of myocardial ischemia or heater probe perforation.

Endoscopic clipping is an emerging modality of endoscopic treatment, it mimics the use of surgical ligature on bleeding artery. Endo-clipping has the theoretical advantage over injection and heater probe in that the tissue reaction or damage will be much milder.

Resolution Clip™ is a newly developed endo-clipping device. It is superior to older generations of endo-clips in that it allows repeated closures and re-opening of clip so as to facilitate accurate deployment onto bleeding artery to ensure its optimal placement for hemostasis.

Consecutive patients with endoscopically confirmed bleeding peptic ulcer will be invited to participate in this double-blind, randomised trial, which compares the efficacy of Resolution clip and conventional dual endoscopic therapy. Patients will be compared for 30-day treatment failure rate.

ELIGIBILITY:
Inclusion Criteria:

* Age >16 , can obtain written consent
* Ulcers that require endoscopic therapy with SRH: Forrest I a, Ib, II a and II b

Exclusion Criteria:

* Moribund patients with terminal malignancy
* Pregnancy
* Intercurrent ulcer complication that prevents treatment and surgery becomes mandatory such as bulbar stenosis and ulcer perforation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Failure to control bleeding endoscopically and recurrent bleeding after initial control | 30 days
  linical rebleeding is defined by fresh hematemesis, fresh melena or hematochezia and signs of hypovolemic shock (systolic blood pressure of <90mmHg and pulse rate >110 per minute) and a drop in hemoglobin of > 2 g/dl per 24 hours despite adequate transfusion.
  Rebleeding will be confirmed by an immediate endoscopy showing fresh blood in stomach or active bleeding from a previously seen ulcer. A clinical rebleeding will be independently reviewed by an adjudication panel.

SECONDARY OUTCOMES:
Transfusion requirement (before and after endoscopic therapy) | within 30 days of therapy
Hospital stay | within 30 days of therapy
The need for surgery | within 30 days of therapy
Mortality from recurrent bleeding and all causes within 30 days of treatment | within 30 days of therapy
Treatment related complications e.g. perforation | within 30 days of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Justin C Wu, MD, Principal Investigator — Endoscopy Center, Prince of Wales Hospital
Locations (1):
- Endocopy Center, Prince of Wales Hospital, Hong Kong SAR, China